CLINICAL TRIAL: NCT07341217
Title: Chemo Brain Prehab Project: Improving Brain Health After Chemotherapy Through Prehabilitation
Brief Title: Chemo Brain Prehab Project
Acronym: CHEMOBRAIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Chris Gaffney (Other)
Responsible Party: Sponsor-Investigator, Dr. Chris Gaffney, Senior Lecturer in Integrative Physiology, Lancaster University
Organization: Lancaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 25/EM/0250; AR2024.07 (Other Grant/Funding Number: North West Cancer Research)
Record Dates: First submitted 2025-12-18; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Older Adults (60 - 85 Years Old); Physically Inactive; Chemotherapy
Keywords: Cancer; Colorectal Cancer; Prehabilitation; Exercise; Brain Health; Chemo-brain; Chemotherapy; Cognitive Function
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Motor Activity | interventions — Geritol; Standard of Care

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation group (Experimental): This group will receive the exercise programme before and during chemotherapy (4 times per week; 2 supervised online home-based sessions and 2 unsupervised home-based sessions), with the addition of daily multivitamins and behavioural support via a weekly telephone check-up.
  Interventions: Behavioral: Exercise Prehabilitation; Dietary Supplement: Multivitamins; Other: Standard Care (in control arm)
- Standard Care Group (Other): This group will receive their treatment as planned as part of standard care, but will not receive the prehabilitation (exercise, nutrition, and behavioural support).
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Behavioral: Exercise Prehabilitation — The prehabilitation group will be asked to undertake a remote exercise programme. The home-based exercise sessions will take place four times per week. Two will be unsupervised exercise sessions, and the other two will be online supervised exercise sessions. Each session will last for approximately 40 minutes for a minimum of 3 weeks, a maximum of 4 weeks. Exercise tolerance will be built up from 2 supervised sessions (week 1) up to the recommended four sessions per week (week 3/4). The number of sessions will be sustained throughout chemotherapy until the end of chemotherapy (visit 3).
  The participants will be remotely supervised by a qualified exercise instructor. They will have a combination of aerobic and resistance exercise within each session. It will be individualised and tailored to their physical abilities. The exercises will target their upper body (arms and shoulders) and legs. Exercise programmes, videos, and links to supervised sessions will be provided.
  Other Names: Exercise programme; exercise intervention
  Arms: Prehabilitation group
Dietary Supplement: Multivitamins — Multivitamins will be given following the first testing visit until the third visit (following the last chemotherapy round). The multivitamins will be taken daily before and during chemotherapy. The multivitamin supplement contains a combination of 24 essential vitamins (vitamin A, D2, B1, B2, B6, B12, C, E, Biotin, nicotinamide, pantothenic acid and folic acid), minerals and trace elements (calcium, iron, copper, phosphorus, magnesium, potassium, zinc, iodine, manganese, selenium, chromium, and molybdenum). Each multivitamin and mineral plays a vital role in the efficient daily maintenance of many body processes.
  Arms: Prehabilitation group
Other: Standard Care (in control arm) — Participants with colorectal cancer will receive chemotherapy treatment.

SUMMARY:
Colorectal cancer is 37% higher in the North West than the national average and is treated by chemotherapy, including fluorouracil, capecitabine, and oxaliplatin. A side effect of these drugs is loss of memory, forgetfulness, and general brain fog, which can persist for months after the end of treatment. These symptoms are collectively known as 'chemo-brain'. An existing prehabilitation intervention that has been previously developed will be used, which increases fitness and reduces hospital length of stay in colorectal cancer surgery patients, to try to improve the symptoms of chemo-brain in those undergoing chemotherapy and improve quality of life.

DETAILED DESCRIPTION:
Colorectal cancer rates in the North West are 37% higher than the national average, with the lowest overall survival in England at 58.1%. Standard chemotherapy drugs such as fluorouracil, capecitabine, and oxaliplatin effectively treat tumours but can damage healthy cells, leading to side effects. One common and distressing effect is known as "chemo-brain", which involves problems with memory, attention, and thinking speed. These symptoms can reduce quality of life and increase stress.

Prehabilitation, which involves exercise and nutritional support before treatment, has demonstrated significant benefits in the surgical setting by improving cardiorespiratory fitness, physical function, and recovery. However, its role before chemotherapy is less clear. Exercise promotes both physical and brain health by increasing growth factors, improving blood flow to the brain, and supporting the formation of new brain cells and blood vessels.

This study aims to investigate whether an exercise-based prehabilitation programme can reduce the symptoms of chemo-brain, improve brain health and enhance quality of life in older adults undergoing chemotherapy for colorectal cancer. Participants aged 60-85 years with stage II or III colorectal cancer scheduled to receive chemotherapy (fluorouracil, capecitabine, or oxaliplatin) are eligible. Suitability to receive chemotherapy must be confirmed by the clinical care team via medical records.

Participants will take part in a remotely supervised exercise programme before and during chemotherapy. The programme consists of four 40-minute sessions per week, including two supervised sessions delivered via video by the lead investigator and two independent sessions supported by an exercise booklet and videos.

Each session includes a warm-up, 20 minutes of aerobic exercise at around 60% of peak fitness, strengthening exercises for upper and lower limbs using resistance bands, and a cool-down. Exercises will be adjusted based on individual ability, with progressions and regressions provided. Participants must have a family member, carer, or friend present during supervised sessions for safety. Psychological support and multivitamin supplementation will also be included.

Assessments will take place at three time points:

* Visit 1 (baseline): 3-4 weeks before chemotherapy.
* Visit 2: Within 72 hours of starting chemotherapy.
* Visit 3: 3-4 days after the final chemotherapy session. A follow-up will occur three months after chemotherapy. At each assessment, cardiorespiratory fitness (CPET), blood samples, brain activity (EEG), cognitive tests, and quality of life questionnaires will be completed.

While there is no guarantee of direct benefit, participation may improve fitness, reduce fatigue, and enhance quality of life during chemotherapy. Exercise can also support mood, manage anxiety and depression, and potentially lessen cognitive changes linked to chemotherapy. Participants will contribute to research that could help improve future cancer care.

Risks are minimal and will be closely managed. CPET carries a small risk of cardiac events or fainting, but all tests will be conducted under medical supervision with appropriate screening, warm-ups, and safety procedures in place. Exercise carries a small risk of muscle strain, but exercises will be tailored to ability.

EEG recordings are safe, though mild skin irritation may occur from the cap or cleaning solution. Blood sampling can cause minor bruising or discomfort, but it will be performed by trained professionals. Cognitive testing may occasionally cause fatigue or frustration.

All procedures will take place in hospital settings with immediate access to medical staff. Any clinical concerns identified during testing will be reported to the participant's oncology team or helpline, following consent procedures. The study will not alter or interfere with normal clinical care.

All data, including personal contact information, will be securely managed within Lancaster University's Microsoft Teams environment, ensuring full GDPR compliance. The study is run by Lancaster University in collaboration with East Lancashire Teaching Hospitals NHS Trust, Lancashire Teaching Hospital NHS Trust, and University Hospitals of Morecambe Bay NHS Trust. Recruitment and testing will take place across all participating sites.

The study is due to begin in early 2026 and will run until September 2027. This study is funded by North West Cancer Research.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with stage II or III colorectal cancer undergoing chemotherapy with fluorouracil, capecitabine, or oxaliplatin.
* Aged 60-85 years old.
* Fluent in English
* Male and female participants
* Not engaged in structured exercise training* within the six months before providing consent.

Exclusion Criteria:

* Presence of comorbidities that may significantly alter the metabolic response to exercise (e.g., diabetes mellitus).
* Current musculoskeletal injury or physical limitations that prevent completion of cardiopulmonary exercise testing (CPET).
* Any contraindication to the multivitamin supplementation (Forceval), including known hypercalcaemia, haemochromatosis, peanut or soya allergy, current use of phenytoin or tetracycline antibiotics, and clinically significant impaired renal or hepatic function.
* Evidence of pre-existing cognitive impairment, including diagnosis of dementia, other neurodegenerative disorders (e.g., Alzheimer's disease), or clinically indicated mild cognitive impairment.
* Diagnosis of atrial fibrillation and haematological malignancy.
* Participants without home internet access will be excluded due to the online delivery of the exercise programme.
* Diagnosis of profound hearing loss.
* Receiving palliative care.
* Presence of synchronous cancer.

  * Structured exercise refers to planned and organised physical activity, such as gym workouts, exercise classes or a team sport, which are designed to improve or maintain physical fitness, often with instruction, rules, and goals.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-09-16 (Estimated); Study Completion 2027-09-16 (Estimated)

PRIMARY OUTCOMES:
Blood-based markers | Blood-based markers will be collected at three visits: baseline (visit 1), 72 hours before the start of chemotherapy (visit 2) and 72 hours after the final dose of chemotherapy has been received (visit 3).
  Use physiological blood-based markers to establish if prehabilitation promotes an improvement in brain health in colorectal cancer patients before starting chemotherapy. Brain-Derived Neurotrophic Factor (BDNF) and Vascular Endothelial Growth Factor (VEGF).
Change in brain activity during the Flanker Inhibitory Control and Attention Test | Data from the Flanker Inhibitory Control and Attention Test will be collected at three visits: baseline (visit 1), 72 hours before the start of chemotherapy (visit 2) and 72 hours after the final dose of chemotherapy has been received (visit 3).
  Cognitive function and its neural correlates will be assessed while participants complete the NIH Toolbox Flanker Inhibitory Control and Attention Test during electroencephalography (EEG) recording. This test assesses inhibitory control and attention by requiring participants to focus on a central target (fish or arrows) and identify its direction while ignoring distracting "flanker" stimuli pointing in a different direction, using a scoring algorithm combining accuracy and reaction time for a cognitive score. Flanker raw scores (0-10) will be converted to age-corrected standard scores (mean 100, standard deviation (SD) 15), with higher scores indicating better cognitive performance. Age-standardised Flanker scores and task-related EEG measures (spectral power ratios and event-related potentials) will be compared across visits 1-3 within participants and between intervention and control groups to examine changes in cognitive performance and associated brain activity.
Change in brain activity during the List Sorting Working Memory Test | Data from the List Sorting Working Memory Test will be collected at three visits: baseline (visit 1), 72 hours before the start of chemotherapy (visit 2) and 72 hours after the final dose of chemotherapy has been received (visit 3).
  Cognitive function and its neural correlates will be assessed while participants complete the NIH Toolbox List Sorting Working Memory Test during electroencephalography (EEG) recording. The test assesses working memory by having individuals recall and sequence visually presented items (such as food and animal pictures) in order of size (smallest to largest) after they disappear. Performance is based on correctly sequenced items. The list sorting raw scores (0-10) will be converted to age-corrected standard scores (mean 100, standard deviation (SD) 15), with higher scores indicating better cognitive performance. Age-standardised list sorting scores and task-related EEG measures (spectral power ratios and event-related potentials) will be compared across visits 1-3 within participants and between intervention and control groups to examine changes in cognitive performance and associated brain activity.
Change in brain activity during the Oral Symbol Digit Test | Data from the Oral Symbol Digit Test will be collected at three visits: baseline (visit 1), 72 hours before the start of chemotherapy (visit 2) and 72 hours after the final dose of chemotherapy has been received (visit 3).
  Cognitive function and its neural correlates will be assessed while participants complete the NIH Toolbox Oral Symbol Digit Test during electroencephalography (EEG) recording. This test is a brief, computerised measure of processing speed, where participants orally match symbols to numbers from a key (1-9) presented on an iPad for 120 seconds, scoring how many correct matches they make sequentially to assess rapid visual information processing. The oral symbol digit raw scores (0-10) will be converted to age-corrected standard scores (mean 100, standard deviation (SD) 15), with higher scores indicating better cognitive performance. Age-standardised oral symbol digit test scores and task-related EEG measures (spectral power ratios and event-related potentials) will be compared across visits 1-3 within participants and between intervention and control groups to examine changes in cognitive performance and associated brain activity.
Changes in brain activity during the Words-In-Noise Test | Data from the Words-In-Noise Test will be collected at three visits: baseline (visit 1), 72 hours before the start of chemotherapy (visit 2) and 72 hours after the final dose of chemotherapy has been received (visit 3).
  Audition and its neural correlates will be assessed while participants complete the NIH Toolbox Words-In-Noise Test during electroencephalography (EEG) recording. The test assesses a person's ability to understand spoken words amidst varying levels of background noise. The test is scored by determining the signal-to-noise ratio (SNR) at which a person correctly repeats 50% of the words, called the SNR50, calculated using the Spearman-Kärber equation. Lower SNR50 values (in dB) indicate better hearing in noise, and higher SNR50 values indicate poorer performance. Participants will be classified as having adequate hearing in noise if their SNR50 is ≤ 6 dB. The SNR50 and task-related EEG measures (spectral power ratios and event-related potentials) will be compared across visits 1-3 within participants and between intervention and control groups to examine changes in cognitive performance and associated brain activity.

SECONDARY OUTCOMES:
Change in Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) total score | The cognitive-related quality of life scores (FACT-Cog) will be collected at three visits: baseline (visit 1) and three months following the final round of chemotherapy.
  The Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) is a self-report questionnaire designed to evaluate how cancer patients perceive their cognitive difficulties, such as memory or concentration issues, and the impact these have on their daily lives and quality of life. The instrument comprises 37 items, each rated on a 5-point Likert scale, yielding a total score ranging from 0 to 148, where higher scores reflect better perceived cognitive functioning and fewer cognitive difficulties. The total FACT-Cog score will be used as the outcome measure to assess change in perceived cognitive function between baseline (before chemotherapy) and three months following the last round of chemotherapy.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - East Lancashire Teaching Hospitals NHS Trust, Blackburn, Lancashire
  - University Hospitals Morecambe Bay Trust, Royal Lancaster Infirmary, Lancaster, Lancashire
  - Lancashire Teaching Hospitals NHS Trust, Preston, Lancashire

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT07341217/Prot_SAP_000.pdf
  • Informed Consent Form (2025-12-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT07341217/ICF_001.pdf